CLINICAL TRIAL: NCT04772417
Title: The Effects of Standardized vs Individualized Seat Height on 1-minute Sit-to-stand Performance
Acronym: ESTI-STS
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02945
Record Dates: First submitted 2021-02-21; First posted 2021-02-26 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Healthy Individuals

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Standardized 1-minute sit-to-stand test — The individuals perform two tests from a standardized chair (seat height 46cm).
Diagnostic Test: Individualized 1-minute sit-to-stand test — The individuals perform two tests from an individualized chair (seat height adjusted so that the starting position elicits a knee flexion angle of 90°).

SUMMARY:
The 1-minute sit-to-stand test (1MSTS) is a widely used functional capacity test and has promising predictive potential. Current standards of practice suggest the use of a chair with a standardized height. However, this practice makes the test more demanding for taller individuals than for shorter individuals. This implies over- or underestimation of functional capacity depending on body morphology.

Therefore, the aim of this study is to investigate the influence of knee joint angle, femur length and bodyweight on the 1MSTS performance in healthy subjects with different morphology.

DETAILED DESCRIPTION:
This is a randomized cross-over trial with the participants performing both procedures twice in one visit. Sufficient breaks in between the tests is granted.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Age 18 and older
* Healthy
* Ability to conduct a 1-minute sit-to-stand-test
* Ability to follow study procedures and instructions in German

Exclusion Criteria:

* Known cardiopulmonary or metabolic diseases (e.g., heart disease, diabetes mellitus etc.)
* Smoking (ex-smoker allowed; if they stopped smoking at least one year before the study inclusion)
* Physical or intellectual impairment precluding informed consent or protocol adherence
* Respiratory infection in the last two weeks
* Pain during sit-to-stand movement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Repetitions in the 1-minute sit-to-stand test | Day 1
  Comparison between the procedures

SECONDARY OUTCOMES:
Predictors towards performance in the 1-minute sit-to-stand test | Day 1
  Comparison between the procedures

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
On reasonable request

REFERENCES:
- [Derived] Kuhn M, Vollenweider S, Clarenbach CF, Kohlbrenner D. The effects of standardised versus individualised seat height on 1-minute sit-to-stand test performance in healthy individuals: a randomised crossover trial. Eur J Appl Physiol. 2023 Jul;123(7):1543-1551. doi: 10.1007/s00421-023-05174-8. Epub 2023 Mar 17. PMID 36932213